CLINICAL TRIAL: NCT03959618
Title: Mono-centric, Prospective, Non-Interventional Study of Quantitative and Qualitative Analysis of Dietary Supplement Taken With Chemotherapy Treatments in Patients With Adjuvant Breast Cancer Taken Care of at the Day Hospital
Brief Title: Intravenous Chemotherapy and Plant-based Dietary Supplements
Acronym: CIVCAP
Status: Completed | Type: Observational
Sponsor: Institut Cancerologie de l'Ouest (Other)
Responsible Party: Sponsor
Other Study IDs: ICO-N-2018-12; 2018-A02460-55 (Registry Identifier: ID RCB)
Record Dates: First submitted 2019-05-15; First posted 2019-05-22 (Actual); Last update posted 2021-05-21 (Actual); Status verified 2021-05

CONDITIONS: Breast Cancer
Keywords: dietary supplements; Desmodium; chemotherapy; breast cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- dietary supplements group: dietary supplements questionary
  Interventions: Other: dietary supplements questionary

INTERVENTIONS:
Other: dietary supplements questionary — Patient Questionary Patient to be carried out at the last cure

SUMMARY:
More and more patients report taking dietary supplements based on herbal medicine, aromatherapy, vitamintherapy,... in the course of their detoxifying anticancer chemotherapy, to stimulate the immune defenses, to relieve and/or decrease the side effects of chemo or even to act against cancer. At European level, there are between 15 and 73% of patients treated for cancer taking a dietary supplement (in particular phytotherapy) or a great heterogeneity according to the studies. However, there is still little evidence of the efficacy of these dietary supplements. A large proportion of patients do not seem to inform their doctor about the use of dietary supplements. Patients using dietary supplements most often ignore the mode of action of these products and generally say they are not informed.

In 2015, at the West Cancerology Institute (ICO), 5 patient files were analyzed taking this type of treatment in addition to chemotherapy; in 2016, 24 files; 2017, 61 patient records and this continues to progress.

At the same time, a product appears very frequently associated with cancer chemotherapy: Desmodium Adscendens, an African plant with in vitro properties of liver protector. The Desmodium contains triterpene saponins, alkaloids, flavonoids, polyphenols, and tryptamine derivatives.

Morevover, several situations of patients undergoing chemotherapy and taking long-term Desmodium, with hepatic cytolyses were experienced, not explained by the usual treatments (case described in the literature).

Therefore, this study will evaluate these new therapeutic modalities that are included in the intake of chemotherapy in order to better know them to improve the therapeutic taking of patients and to focus on the impact of Desmodium in association with chemotherapy.

DETAILED DESCRIPTION:
* Determine the quantitative impact of the use of dietary supplements by patients with breast cancer and treated in a neo-adjuvant and/or adjuvant condition by IV chemotherapy in day hospital.
* Determine an over-risk of disruption of liver balance in the population of patients taking Desmodium.
* Gather a critical mass of relevant information with the objective of carrying out the evaluation and analysis of cancer care practices related to the intake of dietary supplements.

ELIGIBILITY:
Inclusion Criteria:

* breast cancer treated by intra-venous chemotherapy
* inclusion at the last cycle (cure)
* all chemotherapy cycles realised at ICO

Exclusion Criteria:

* no breast cancer
* metastatic breast cancer
* not all chemotherapy cycles realised at ICO
* patient who has not finished his chemotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients of the ICO René Gauducheau taken care at day hospital for IV chemotherapy treatment of breast cancer in neoadjuvant and/or adjuvant situation.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2019-04-02 (Actual); Primary Completion 2020-05-13 (Actual); Study Completion 2020-05-13 (Actual)

PRIMARY OUTCOMES:
evaluate quantitatively the use of dietary supplements in patients during IV chemotherapy | 12 months
  rate of patients taking a dietary supplement

SECONDARY OUTCOMES:
Evaluate the impact of taking Desmodium between the first and last cycle of treatment | 12 months
  % of patients with hepatic cytolysis undergoing chemotherapy between the first and last treatments
Description of dietary supplements taken | 12 months
  Description of different types of dietary supplements

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuelle BOURBOULOUX, MD, Principal Investigator — ICO
Locations (1):
- Institut de Cancerologie de L'Ouest, Saint-Herblain, France